CLINICAL TRIAL: NCT06708533
Title: Investigating the Gut Microbiome and Symptomology in IBS: Mechanisms and Therapeutic Implications for Symptom Relief Through Prescribed Physical Activity in Clinical Practice
Brief Title: Investigating the Gut Microbiome and Symptomology in IBS
Acronym: MICROFIT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nottingham Trent University (Other)
Collaborators: Nottingham University Hospitals NHS Trust (Other); University of Reading (Other)
Responsible Party: Principal Investigator, Hannah Lindsell, Ms, Nottingham Trent University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 345554
Record Dates: First submitted 2024-11-21; First posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Irritable Bowel Syndrome (IBS)
Keywords: Physical Activity; Irritable Bowel Syndrome; Gut Microbiome; Exercise; IBS
MeSH Terms: conditions — Irritable Bowel Syndrome; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 12-week physical activity programme (Experimental): Participants in this arm will engage in a structured 12-week walking program. They will complete sub-maximal fitness assessments and provide biological samples during visits to the university at baseline, week 6, and week 12. They will also complete questionnaires assessing IBS symptoms, quality of life (QoL), anxiety, depression, and other factors.
  Interventions: Behavioral: Physical Activity
- No intervention control group (No Intervention): Participants in this arm will not receive any intervention and will continue their usual lifestyle for the study duration. They will complete the same assessments as the intervention arm, including providing biological samples, undergoing sub-maximal fitness tests, and completing questionnaires at baseline, week 6, and week 12. This arm serves as a comparison group to evaluate the effects of the walking program.

INTERVENTIONS:
Behavioral: Physical Activity — This intervention involves a structured 12-week walking program designed to increase routine physical activity among participants diagnosed with IBS. The intervention focuses on moderate-intensity walking, performed regularly, in line with World Health Organisation (WHO) guidelines with the aim of relieving IBS symptoms.
  Key elements include:
  Participants will be guided to adhere to an individualised walking protocol, ensuring consistency in activity levels.
  Physical activity levels will be monitored using self-reported diaries and wearable activity trackers to ensure compliance.
  Participants will also attend three scheduled visits to the university (baseline, week 6, and week 12) for biological sample collection, sub-maximal fitness assessments, and the completion of validated questionnaires on IBS symptoms, quality of life (QoL), anxiety, and depression.
  Arms: 12-week physical activity programme

SUMMARY:
This intervention study explores whether a routine physical activity intervention can help manage or relieve symptoms of Irritable Bowel Syndrome (IBS) in adults who have been clinically diagnosed with IBS. The main questions it aims to answer is:

• Primary Outcome: Does engaging in routine physical activity reduce the severity of IBS symptoms compared to baseline levels?

Comparison Group: Researchers will compare the intervention group (receiving the 12-week physical activity program) with a control group (receiving no intervention for 12-weeks).

Participant Activities and Interventions:

* Complete a 12-week walking programme.
* Visit the university on 3 occasions (baseline, week-6 and week-12) for biological sample collection and sub-maximal fitness assessments.
* Complete a series of subjective health related questionnaires.

DETAILED DESCRIPTION:
This study investigates the effects of a structured routine physical activity intervention on symptom management in adults with irritable bowel syndrome (IBS). The intervention consists of a 12-week walking program designed to assess whether regular physical activity can reduce IBS symptom severity and improve quality of life.

Participants are assigned to either the intervention group, where they will engage in routine walking sessions, or to a control group, which will not participate in the physical activity program. The primary outcome is the reduction in IBS symptom severity compared to baseline, with secondary outcomes including quality of life (QoL) scores, anxiety, and depression levels in addition to biological markers.

Study activities include:

* Walking Program: Participants in the intervention group will follow a personalised moderate-intensity walking program, with frequency and duration tailored to meet a 12-week schedule and personalised to individual 6-minute walk test results.
* University Visits: All participants will attend three university visits at baseline, week 6, and week 12. During these visits, biological samples will be collected for the assessment of gut microbiome, metabolome, proteome, and sub-maximal fitness assessments (6-minute walk test and hand grip strength) will be conducted.
* Questionnaires: Participants will complete validated questionnaires assessing IBS symptoms, quality of life, and psychological well-being (including anxiety and depression) at each visit to track any changes over time.

The study aims to provide insights into the potential benefits of physical activity as a non-pharmacological management strategy for IBS management.

ELIGIBILITY:
Inclusion Criteria:

* Be 18-64 years old
* Have CLINCALLY DIAGNOSED IBS
* Know your IBS-SUBTYPE (e.g., constipation, diarrhoea, mixed/alternating)

Exclusion Criteria:

* Pregnant or breastfeeding
* Organic gastrointestinal conditions (Inflammatory Bowel Disease, Coeliac Disease, Colorectal Cancer)
* On medication with known influence on gastrointestinal motility (thyroid disease, diabetes mellitus, coeliac disease and neurological disease)
* Have used antibiotics in the past 3 months
* Currently using opioid pain medications (except occasional/non-daily use of NSAIDs)
* Regular consumption of pre- and probiotic foods/supplements
* Completing more than 300-minutes of PA per week

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Clinically significant change in IBS Symptom Severity Score (IBS-SSS) | Baseline, Week 6, Week 12
  The primary outcome will assess changes in IBS symptom severity over the 12-week intervention using a validated measure such as the IBS Severity Scoring System (IBS-SSS). This includes self-reported symptom scores for pain, frequency of bowel disturbances, and overall impact on daily life.
  A scale of 0-500, with higher scores indicative of more severe symtpoms and a change in 50points indicates a clinically significant change.
  The categories:
  Healthy: 0-74 Mild IBS: 75 ≤ Score < 175 Moderate IBS: 175 ≤ Score < 300 Severe IBS: Score ≥ 300

SECONDARY OUTCOMES:
Changes in Gut Microbiota Composition | Baseline, Week 6, Week 12
  Biological samples (e.g., stool) will be analysed to assess changes in gut microbiota composition. This aims to elucidate potential mechanisms underlying symptom relief associated with the intervention. Specific analyses will include:
  - Characterisation of microbial diversity and abundance using next-generation sequencing (e.g., 16S rRNA sequencing).
Changes in Metabolomic Profiles | Baseline, Week 6, Week 12
  Biological samples (e.g., blood) will be analysed to assess changes in metabolomic profile. This aims to elucidate potential mechanisms underlying symptom relief associated with the intervention. Specific analyses will include:
  - Identification of key metabolites and pathways involved through untargeted metabolomics.
Changes in Proteome | Baseline, Week 6, Week 12
  Biological samples (e.g., blood) will be analysed to assess changes in gut proteome profile. This aims to elucidate potential mechanisms underlying symptom relief associated with the intervention. Specific analyses will include:
  - Proteomic analysis to explore systemic changes and molecular signatures linked to IBS symptom modulation.
Physical Fitness Improvement | Baseline, Week 6, Week 12
  Sub-maximal fitness tests will assess changes in participants' aerobic capacity as an indicator of physical activity levels.
Changes in Anxiety Levels | Baseline, Week 6, Week 12
  Evaluated using the Generalized Anxiety Disorder-7 (GAD-7) self report questionnaires.
  Participants rate how often they've experienced seven symptoms over the past two weeks, with each item scored from 0 ("Not at all") to 3 ("Nearly every day").
  The total score is calculated by summing the responses, with a maximum score of 21. Higher scores indicate greater anxiety severity, categorised as follows:
  None: 0-4 Mild: 5-9 Moderate: 10-14 Severe: 15-21
Changes in Depression Levels | Baseline, Week 6, Week 12
  Evaluated using the Patient Health Questionnaire-8 (PHQ-8) self report questionnaires.
  Participants rate how often they've experienced eight symptoms over the past two weeks, with each item scored from 0 ("Not at all") to 3 ("Nearly every day").
  The total score is the sum of responses, with a maximum score of 24. Higher scores indicate greater depression severity, categorised as follows:
  None: 0-4 Mild: 5-9 Moderate: 10-14 Moderately Severe: 15-19 Severe: 20-24
Change in Quality of Life (QoL) Scores | Baseline, Week 6, Week 12
  Assessed using a validated Short Form Health Survey (SF-36), QoL questionnaire.
  The SF-36 is a health survey assessing quality of life across 9 domains:
  Physical Functioning, Role Limitations due to Physical Health, Role Limitations due to Emotional Health, Energy/Fatigue, Emotional Well-Being, Social Functioning, Pain, General Health, and Health Change.
  Each domain is scored from 0 to 100, with higher scores indicating better health.